CLINICAL TRIAL: NCT05643131
Title: Evaluation of the Hyivy Device as a Non-hormonal Therapy in People With Endometriosis
Brief Title: Hyivy Device as Non-hormonal Therapy in Endometriosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyivy Health Inc (Industry)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYV-001-C23
Record Dates: First submitted 2022-08-18; First posted 2022-12-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Endometriosis; Pelvic Pain; Dilator
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Prospective observational pre/post repeated-measures pilot intervention study
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyivy Intravaginal Device (Experimental): Participants will receive a Hyivy intravaginal device for at-home use. Recommended use is three times per week for 12 weeks and consists of 10 minutes of heat (37-39ºC) and 10 minutes of dilation per session.
  Interventions: Device: Hyivy Intravaginal Device

INTERVENTIONS:
Device: Hyivy Intravaginal Device — Intravaginal use of Hyivy device three times per week for 12 weeks, with each session consisting of 10 minutes of heat (37-39ºC) and 10 minutes of dilation.

SUMMARY:
This study seeks to address accessible management of endometriosis-associated chronic pelvic pain by evaluating a novel device used in the home. The study is designed as a proof-of-concept single-arm pilot study, and the primary objective is to assess change in overall self-reported pelvic pain in people with endometriosis-associated chronic pelvic pain following the use of the Hyivy intravaginal device.

DETAILED DESCRIPTION:
Endometriosis is a chronic, inflammatory, estrogen-dependent disease characterized by ectopic growth of uterine-like cells outside the uterus. People living with endometriosis typically experience debilitating pelvic pain (dysmenorrhea, dyspareunia, dyschezia, dysuria, non-menstrual pelvic pain), and infertility. Endometriosis also has significant negative impacts on quality of life, physical, mental, and social wellbeing.

There is no diagnostic marker nor cure for this chronic disease. Current treatment options include medical therapies (mainly hormonal treatments aimed at suppressing menstruation or growth of the ectopic cells), surgery (to remove endometriotic lesions/nodules), and complementary or alternative therapies (non-medical or surgical options to manage symptoms; heat, mindfulness, diet, yoga, natural remedies, physical therapies, etc.).

Many people living with endometriosis report having used self-management strategies (complementary and alternative therapies) to manage their symptoms, and research on treatments and alternative therapies are consistently ranked among the top endometriosis research priorities. Alternative therapies have the potential to complement existing medical and surgical therapies, offering additional options to manage symptoms like pain.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 at the time of enrollment
* 2.Generally in good health (other than due to endometriosis), at physician's discretion
* 3.Diagnosed with endometriosis (clinical, radiologic, or surgical)
* 4.Diagnosed with chronic pelvic pain (self-reported pain in pelvic area lasting >3 months)
* 5.VAS for overall pelvic pain ≥ 4 at screening and baseline
* 6.Medically managing endometriosis using continuous hormonal medications (i.e., oral contraceptive pills, progesterone only pills, Mirena, GnRH agonists/antagonists) for at least 3 months prior to enrollment
* 7.Agrees not to commence any new treatments (medical or physical therapies) for the 12-week intervention period, including hormonal therapies for any medical condition, and complimentary and/or alternative management of surgery for endometriosis and associated chronic pain
* 8.Agrees not to undergo pelvic physiotherapy with a trained professional during the study
* 9.Agrees to avoid taking non-steroidal anti-inflammatory drugs (e.g., ibuprofen) for 72 hours before Visits 1, 2, and 3
* 10.Must have the ability to charge the investigational device
* 11.Must be willing and able to insert intravaginal device
* 12.Able to understand, comply and consent to protocol requirements and instructions
* 13.Able to attend scheduled study visits and complete required investigations

Exclusion Criteria:

* 1.Chronic pelvic pain thought to be due to a condition other than endometriosis
* 2.Diagnosis of premature ovarian insufficiency
* 3.Any other medical condition or clinical finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational product or that may affect the interpretation of the results or leave the patient at high risk from treatment complications, at the discretion of the investigator(s)
* 4.Any surgery in the past 3 months or anticipates having surgery during the study
* 5.Allergy to Hyivy device's materials
* 6.Active vaginal infection (e.g. vulvovaginal candidiasis, trichomonas vaginitis, bacterial vaginosis, STIs) or infection in the pelvic area
* 7.Current use of antibiotics and a history of vulvovaginal candidiasis
* 8.Pregnant or lactating
* 9.Currently under the care of a pelvic floor physiotherapist
* 10.Have open wounds, cuts, or open sores present in vaginal or pelvic area
* 11.Severe atrophic vaginitis or very dry, itchy, or sore vagina/vaginal area, at the discretion of the primary investigator(s)
* 12.Hypoesthesia or loss in sensation of the pelvic floor
* 13.Total and/or partial prolapse of the uterus and/or vagina
* 14.Symptoms of severe urinary retention, severe extra-urethral incontinence or overflow incontinence
* 15.Unable to position the device according to directions for use
* 16.Use of any medical devices that may interfere with the investigational device's function, such as pacemakers, ventilators, and ear implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall self-reported pelvic pain | Baseline, 6-weeks, 12-weeks
  Overall pelvic pain will be evaluated using a digital visual analog scale (VAS)

SECONDARY OUTCOMES:
Site-specific tenderness and pelvic floor muscle pain | Baseline, 6-weeks, 12-weeks
  Site-specific tenderness and pelvic floor muscle pain will be measured by the Biberoglu and Behrman scale (B&B) ranging from 0 (none) to 15 (severe) and patient exams
Quality of Life (EHP-30) | Baseline, 6-weeks, 12-weeks
  Changes in quality of life as assessed by the Endometriosis Health Profile-30 (EHP-30) ranging from 0 (best possible health status) to 100 (worst possible health status).
Sexual Function (FSFI) | Baseline, 6-weeks, 12-weeks
  Changes in sexual function as assessed by the Female Sexual Function Index (FSFI). Scores range from 2 to 36 with higher scores indicating greater functioning.
Safety and tolerability of the Hyivy device | Up to 12-weeks
  Occurrence of adverse events (AE) and serious adverse events (SAE).
Adherence to study protocol | 6-weeks, 12-weeks
  Usage data collected by the Hyivy device will be used to assess participant adherence to the study regimen of 3 times/week device use.
Feasibility of the Hyivy device | 6-weeks, 12-weeks
  Device usage will be assessed with a study-specific questionnaire.
Use of rescue medication | Baseline, 6-weeks, 12-weeks
  Changes in the use of rescue medications for chronic pelvic pain, assessed with a study-specific questionnaire.

OTHER OUTCOMES:
Autonomic function | Baseline, 6-weeks, 12-weeks
  Autonomic nervous system (ANS) function will be assessed using measures of heart rate variability (HRV) during a deep breathing test, active standing test, and water intake test.
Peripheral gene expression | Baseline, 6-weeks, 12-weeks
  Changes in peripheral inflammation as assessed by a protein biomarker panel before and after device use
Emergency room (ER) visits | Baseline, 6-weeks, 12-weeks
  Number of ER visits due to chronic pelvic pain in the last 6 weeks
Device usability and patient satisfaction | 12-weeks
  Study-specific questionnaire to gather patient feedback

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Leonardi, M.D., Principal Investigator — McMaster University Medical Centre
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Singh S, Soliman AM, Rahal Y, Robert C, Defoy I, Nisbet P, Leyland N. Prevalence, Symptomatic Burden, and Diagnosis of Endometriosis in Canada: Cross-Sectional Survey of 30 000 Women. J Obstet Gynaecol Can. 2020 Jul;42(7):829-838. doi: 10.1016/j.jogc.2019.10.038. Epub 2020 Jan 27. PMID 32001176
- [Background] Kong S, Zhang YH, Liu CF, Tsui I, Guo Y, Ai BB, Han FJ. The complementary and alternative medicine for endometriosis: a review of utilization and mechanism. Evid Based Complement Alternat Med. 2014;2014:146383. doi: 10.1155/2014/146383. Epub 2014 Feb 19. PMID 24701237
- [Background] Vercellini P, Vigano P, Somigliana E, Fedele L. Endometriosis: pathogenesis and treatment. Nat Rev Endocrinol. 2014 May;10(5):261-75. doi: 10.1038/nrendo.2013.255. Epub 2013 Dec 24. PMID 24366116
- [Background] Becker CM, Gattrell WT, Gude K, Singh SS. Reevaluating response and failure of medical treatment of endometriosis: a systematic review. Fertil Steril. 2017 Jul;108(1):125-136. doi: 10.1016/j.fertnstert.2017.05.004. PMID 28668150
- [Background] As-Sanie S, Black R, Giudice LC, Gray Valbrun T, Gupta J, Jones B, Laufer MR, Milspaw AT, Missmer SA, Norman A, Taylor RN, Wallace K, Williams Z, Yong PJ, Nebel RA. Assessing research gaps and unmet needs in endometriosis. Am J Obstet Gynecol. 2019 Aug;221(2):86-94. doi: 10.1016/j.ajog.2019.02.033. Epub 2019 Feb 18. PMID 30790565
- [Background] Duffy J, Hirsch M, Vercoe M, Abbott J, Barker C, Collura B, Drake R, Evers J, Hickey M, Horne AW, Hull ML, Kolekar S, Lensen S, Johnson NP, Mahajan V, Mol BW, Otter AS, Puscasiu L, Rodriguez MB, Rombauts L, Vail A, Wang R, Farquhar CM; endo:outcomes - an International Collaboration Harmonising Outcomes and Outcome Measures for Endometriosis Research. A core outcome set for future endometriosis research: an international consensus development study. BJOG. 2020 Jul;127(8):967-974. doi: 10.1111/1471-0528.16157. Epub 2020 Mar 30. PMID 32227676
- [Background] Nnoaham KE, Hummelshoj L, Webster P, d'Hooghe T, de Cicco Nardone F, de Cicco Nardone C, Jenkinson C, Kennedy SH, Zondervan KT; World Endometriosis Research Foundation Global Study of Women's Health consortium. Impact of endometriosis on quality of life and work productivity: a multicenter study across ten countries. Fertil Steril. 2011 Aug;96(2):366-373.e8. doi: 10.1016/j.fertnstert.2011.05.090. Epub 2011 Jun 30. PMID 21718982